CLINICAL TRIAL: NCT01654822
Title: Single Center, Placebo Controlled, Double-Blind Study to the Treatment of HPV Infected Cervix With AV2 Antiviral Spray and Assessment of Viral Load
Brief Title: AV2 Antiviral Spray Versus Placebo in Human Papillomavirus Cervix Infections
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cesa Projects International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AV2-HPV-001
Record Dates: First submitted 2012-06-19; First posted 2012-08-01 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Genital Human Papilloma Virus Infection
Keywords: HPV; cervix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- olive oil with 10% d-limonene (Placebo Comparator): Topical spray one-time administration 2 puffs of 100µl
  Interventions: Drug: topical spray on the cervix; Procedure: cervical swab with Cervex-Brush-Combi at T0; Procedure: cervical swab with Cervex-Brush-Combi at T1
- AV2-DM antiviral spray (Experimental): Topical spray one-time application 2 puffs of 100µl
  Interventions: Drug: topical application cervical spray; Procedure: cervical swab with Cervex-Brush-Combi at T0; Procedure: cervical swab with Cervex-Brush-Combi at T1

INTERVENTIONS:
Drug: topical application cervical spray — one time (2 puffs) topical application of 100µl AV2-DM antiviral spray( containing 50% AV2-DM and 50% olive oil)on the cervix
  Arms: AV2-DM antiviral spray
Drug: topical spray on the cervix — one time (2 puffs) topical spray of 100 µl (90% olive oil and 10% d-limonene) on the cervix
  Arms: olive oil with 10% d-limonene
Procedure: cervical swab with Cervex-Brush-Combi at T0
  Arms: AV2-DM antiviral spray
Procedure: cervical swab with Cervex-Brush-Combi at T1
  Arms: AV2-DM antiviral spray
Procedure: cervical swab with Cervex-Brush-Combi at T0
  Arms: olive oil with 10% d-limonene
Procedure: cervical swab with Cervex-Brush-Combi at T1
  Arms: olive oil with 10% d-limonene

SUMMARY:
This study aims to prove that, by a one-time topical spray on the cervix, AV2-DM is an effective antiviral in reducing on short term (3 months) the human papillomavirus (HPV) infection.

* Primary endpoint: significant drop in viral load AV2-DM versus placebo
* Secondary endpoint:the number of patients with adverse events

ELIGIBILITY:
Inclusion Criteria:

1. Women between 25 and 40 years
2. Patient has been recently (up to 6 months) Quantitatively (Viral Load) and Qualitatively (HPV types) diagnosed with HPV.
3. Ability and willingness to participate in the study.
4. Subject agrees to refrain from using prescription or supplemental antiviral medications without obtaining permission of the Treating Doctor.
5. Voluntary written informed consent.

Exclusion Criteria:

1. Subject has been vaccinated against HPV
2. Interval between a delivery and T0 is less than 3 months
3. Subject has a gynecologic surgical intervention between T0 and T1
4. Subject is diagnosed HPV negative at T0
5. Subject has a (adeno)carcinoma in situ.
6. Females with child bearing potential who are not using a reliable, medically accepted method of birth control
7. Pregnant or breast-feeding female, or women planning to become pregnant during the trial.
8. Medical history of immunosuppression by radiotherapy, chemotherapy, immuno-modulatory drugs, or HIV.
9. Participation to another clinical trial concerning HPV infections within 6 months before the application of AV2-DM antiviral spray.
10. Medical history of any severe diseases like hepatitis, renal or liver dysfunction, car-diovascular, gastrointestinal, malignant tumor(s), or psychiatric disorders etc., which might influence the assessments or conduct of the trial by the discretion of the investigator.
11. Intake or application of antivirals or other prohibited concomitant medication within 30 days prior to application of AV2, or patients who plan to take such drugs during the trial.
12. Known or suspected allergic or adverse response to the investigational product AV2-DM Antiviral spray, it's components, olive oil or d-limonene.
13. Inability to follow the study protocol.

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-08; Primary Completion 2012-12 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy comparison number of patients with drop (min 2 Log units) in HPV specific viral load AV2-DM versus placebo | 90 days

SECONDARY OUTCOMES:
number of adverse vents AV2-DM versus placebo | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Labo Riatol, Antwerp, Antwerpen, Belgium